CLINICAL TRIAL: NCT04731623
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending, Dose-Escalation, Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ION904 Administered Subcutaneously to Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ION904
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION904-CS1
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Participants; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ION904 (Experimental): Single ascending dose of ION904 will be administered by SC injection on Day 1.
  Interventions: Drug: ION904
- Placebo (Placebo Comparator): Placebo (0.9% sterile saline) will be administered by SC injection on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ION904 — ION904 will be administered by SC injection.
  Arms: ION904
Drug: Placebo — Placebo (0.9% sterile saline) will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ION904.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-ascending dose escalation study of ION904 in up to 72 participants. Following a Screening Period of up to 28 days, eligible healthy participants will be randomized to treatment and receive a single, subcutaneous (SC) dose of the assigned study drug. Participants will be followed for up to 13 weeks after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Must be healthy males, or females of non-childbearing potential, aged 18 to 65 at the time of informed consent
2. Females must be either surgically sterile or post-menopausal; males must be abstinent, surgically sterile, or if engaged in sexual relations with a woman of childbearing potential, a highly effective contraceptive method must be used from the time of signing the informed consent form until at least 13 weeks after the last dose of Study Drug or the healthy participant must be abstinent through this time period
3. Willing to refrain from strenuous exercise/activity (for example heavy lifting, weight training, intense aerobics classes etc.) for at least 24 hours prior to study visits
4. Body mass index (BMI) requirements between 18 and 35 kg/m^2

Exclusion Criteria:

1. Clinically significant abnormalities in medical history or physical examination
2. Uncontrolled arterial hypertension
3. Active infection with human immunodeficiency virus (HIV), hepatitis C or hepatitis B or prior treatment for hepatitis C
4. Treatment with another investigational drug, biological agent, or device within 1 month of Screening
5. History of bleeding diathesis or coagulopathy
6. Regular use of alcohol within 6 months prior to screening, or use of soft drugs within 3 months prior to Screening, or hard drugs within 1 year prior to Screening, or positive urine drug screen at Screening
7. History of any severe (e.g., anaphylaxis) drug allergies
8. History of hypersensitivity to other antisense oligonucleotides (ASOs)
9. Concomitant medication restrictions: over-the-counter or prescription medications within 14 days, prior to dosing on Day 1. Accepted exceptions are:

   * Acetaminophen (paracetamol) up to 2 grams per day (g/d) or ibuprofen up to 2.4 g/day taken sporadically for analgesia
   * Thyroid hormone replacement therapy provided participant is stable on replacement therapy (and participant is euthyroid)
   * Other possible exceptions must be reviewed and acknowledged by the Investigator in consultation with Sponsor's Medical Monitor
10. Blood donation of 50 to 499 mL within 30 days of Screening or of > 499 mL within 60 days of Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) | Up to Day 85
Severity and dose relationship of TEAE | Up to Day 85
Severity and dose relationship of clinically significant changes in laboratory values | Up to Day 85
Severity and dose relationship of clinically significant changes in ECG | Up to Day 85

SECONDARY OUTCOMES:
Changes in the Level of ION904 Target Biomarker | Up to Day 85
Cmax: Maximum Observed Plasma Concentration of ION904 | Up to Day 85
Tmax: Time to Reach the Maximum Plasma Concentration of ION904 | Up to Day 85
t½λz: Plasma Elimination Half-life of ION904 | Up to Day 85
AUC0-t: Area Under the Plasma Concentration-Time Curve from Time Zero to Time t for ION904 | Up to Day 85
Urine 0-24 Hour (hr) Excretion of ION904 | Up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- BioPharma Services, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No